CLINICAL TRIAL: NCT05739773
Title: Evaluation of the Effect of Five Elements Music Combined With Binaural Beat on Sleep Disorder
Brief Title: Evaluation of the Effect of Combined Music on Sleep Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Yueh-Ting Tsai, Assistant professor, China Medical University, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P11001; CMUH110-REC1-170 (Other: ChinaMUH)
Record Dates: First submitted 2022-11-05; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): the five-element music group
  Interventions: Other: five-element music therapy
- Control (Placebo Comparator): binaural beats group
  Interventions: Other: five-element music therapy

INTERVENTIONS:
Other: five-element music therapy — music therapy
  Other Names: binaural beats

SUMMARY:
The results of this study will provide an affordable, safe and scientific treatment for patients with sleep disorders, so that patients can improve their sleep quality at home.

DETAILED DESCRIPTION:
The population suffered from sleep disorders is raising year by year, it has increased much social costs and medical burdens, especially the spread of the COVID-19 epidemic has made it even worse recently. Although many studies in the past few years have found that the use of non-invasive music therapy (such as five-element music, music combined with binaural beats) can effectively improve sleep quality, however, there is a lack of rigorous study design and measurement tools (scientific instrument examination).

To explore the effects of short-term sleep quality in patients with sleep disorders after receiving five-element music therapy or binaural beats, and further explore the combination of the above two music therapies to verify its effectiveness in improving long-term sleep quality.

The first year study was a randomized single-blind trial. 60 patients with sleep disorders were randomly assigned to the five-element music group and binaural beats group for two consecutive nights treatment to verify their short-term effects and assess the differences between them; the second year study was a randomized controlled trial , 60 patients with sleep disorders were randomly assigned to the five-element music combined with binaural beats group and the control group for four-week follow-up treatment to verify their long-term results and evaluate the feasibility of home treatment. The main results were measured with meridian energy examination and polysomnography. Other secondary results include sleep-related questionnaires (including Pittsburgh Sleep Quality Index, Epworth Sleepiness Scale, Berlin Questionnaire, Hospital Anxiety and Depression Scale).

ELIGIBILITY:
Inclusion Criteria:

* sleep disorder
* PSQI score > 5

Exclusion Criteria:

* Using tranquilizers or taking drugs or foods (such as coffee or refreshing drinks)
* Severe cardiopulmonary disease (heart failure or cardiopulmonary failure) or cancer
* Kidney dialysis patients
* Patients with cardiac rhythm regulators or built-in hearing aids
* Pregnant women and women who are still breastfeeding

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-08-11 (Estimated); Study Completion 2023-10-11 (Estimated)

PRIMARY OUTCOMES:
polysomnography | two consecutive nights
  Polysomnography refers to a systematic process used to collect physiologic parameters during sleep
change meridian energy | two consecutive nights
  Meridian energy examination

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | two consecutive nights
  sleep-related questionnaire
Epworth Sleepiness Scale | two consecutive nights
  sleep-related questionnaire
Berlin Questionnaire | two consecutive nights
  sleep-related questionnaire
Hospital Anxiety and Depression Scale | two consecutive nights
  sleep-related questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Ting Tsai, Principal Investigator — China Medical University, Taiwan
Locations (1):
- Yueh-Ting Tsai, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No